CLINICAL TRIAL: NCT04939493
Title: Use of Rhythmic Auditory Cueing During Bilateral Training of the Upper Extremities in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Hesham Mohamed Abdelhady, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Reem_MSc
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Hemiplegia, Spastic
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhythmic Auditory Cueing (Experimental): Group (B): Patients in this group will receive the same designed physical therapy program given to the control group in addition to auditory cueing during bilateral arm training using the metronome.
  Interventions: Other: Rhythmic Auditory Cueing; Other: Bilateral arm training; Other: Conventional physical therapy program
- Bilateral arm training (Active Comparator): Patients in this group will receive a standard physical therapy program in addition to Bilateral arm training.
  Interventions: Other: Bilateral arm training; Other: Conventional physical therapy program

INTERVENTIONS:
Other: Rhythmic Auditory Cueing — Patients will perform the same movement sequence in time with the metronome beat. The frequency of the rhythmic auditory stimulation will be matched to the participant"s preferred movement speed, which will be assessed prior to the start of the trial, and participants typically started moving after they had heard the metronome beat two to three times. Participants will be given sufficient practice trials to ensure full understanding before the actual recording of data, and will be given 3-minutes break between trials.
  On the 3rd and 5th week, the rhythm frequency was increased by 5%.
  Arms: Rhythmic Auditory Cueing
Other: Bilateral arm training — Training will consist of 20 minutes of bilateral arm training In each session, patients will be seated comfortably at a table in the following limb positions: ankles in neutral dorsiflexion, knees and hips placed at 90°, shoulders in 0° flexion, elbows in 60° flexion, and wrists in neutral position of flexion/extension
Other: Conventional physical therapy program — Scapular mobilization. Thoracic spine mobilization. Mechanical assisted (active and passive) exercises. Therapeutic positioning as weight bearing on the paretic arm. Opening and closing closed fist. Strengthening exercise. Stretching of spastic muscles.

SUMMARY:
The purpose of the study is to determine the effect of rhythmic auditory cueing with bilateral arm training on upper limb functions in stroke patients.

DETAILED DESCRIPTION:
Arm and hand movement problems are major contributors to disability in patients after stroke. In fact, only 5% of adults regain full arm function after stroke, and 20% regain no functional use. Hence, alternative strategies are needed to reduce the long-term disability and functional impairment from upper limb hemiparesis.

To solve problems concerning upper limb dysfunction related to stroke, various treatment methods have been used in several previous studies. Rhythmic auditory stimulation has been reported as an effective intervention for improving movement in the affected extremities of stroke patients.

To the best of our knowledge, no mentioned previous studies evaluating the effect of rhythmic auditory cueing with bilateral arm training using functional exercises on upper extremity impairment in patients with stroke in Egypt are reported. So, this study aims to determine the effect of rhythmic auditory cueing with bilateral arm training on upper limb functions in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Thirty patients with ischemic stroke from both sexes will be included.
2. Patients will have stroke for the first time.
3. The age of patients will range from 45 to 60 years.
4. Duration of illness will be from six months to eighteen months.
5. The degree of spasticity will ranged from 1 to 1 + grade according to the modified Ashworth scale.
6. Patients will have moderate arm motor impairment (between 30 and 49 scores) according to Fugl-Meyer (FM) arm section scale.
7. The affected upper extremity will be the dominant side.
8. Patients will be able to sit and maintain balance in a sitting position.

Exclusion Criteria:

* The patients will be excluded if they have:

  1. Visual or auditory deficits.
  2. Perceptual disorders.
  3. Any surgical interventions in the upper extremities limiting the range of motion.
  4. Aphasia or apraxia.
  5. Musculoskeletal or neurological impairment of the unaffected upper extremity.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Assessing the change in Upper Extremity Motor Performance | Baseline and 6 weeks post-intervention
  Assessment via using Upper Extremity Motor Performance scale. This scale has been shown to be valid and reliable, and it correlates well with inter joint upper extremity coordination. It has a maximum score of 66
Assessing the change in upper limb Motor Function | Baseline and 6 weeks post-intervention
  Assessment via using Wolf Motor Function Test (WMFT) The final time score will be the median time required for all timed tasks executed. One hundred twenty seconds is the maximum time allowed for each task attempted Timing is carried out using a stopwatch.
Assessing the change in gross manual dexterity | Baseline and 6 weeks post-intervention
  Assessment via using Box and Block Test Involves moving 1-inch cube blocks from a rectangular box container to another container, and the number of blocks moved by each hand in 60 seconds is determined using stop watch

CONTACTS AND LOCATIONS:
Overall Officials: Reem Abdelhady, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic - Faculty of Physical Therapy - Cairo University, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No